CLINICAL TRIAL: NCT07056673
Title: Efficacy and Safety of Cold Atmospheric Plasma for Moderate-to-severe Acne Vulgaris: a Multicentre, Randomised, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Cold Atmospheric Plasma for Moderate-to-severe Acne Vulgaris Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: the 989th Hospital of Chinese People's Liberation Army Joint Logistic Support Force (Unknown)
Responsible Party: Principal Investigator, Lin Tao, MM, Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAP630
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Cold atmospheric plasma
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: For the placebo group, the device will be operated with the plasma-generating field disabled, so that no plasma will be produced. Only environmental cues such as sound will be simulated to ensure blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the CAP treatment group (Active Comparator)
  Interventions: Device: Active CAP therapy; Other: standard care based on the JAAD acne guidelines
- the placebo group (Placebo Comparator)
  Interventions: Device: sham CAP therapy; Other: standard care based on the JAAD acne guidelines

INTERVENTIONS:
Device: Active CAP therapy — The patients in the CAP group will receive six sessions of CAP treatment, administered once weekly for six consecutive weeks. If complete clearance of facial acne is achieved before all six sessions, CAP treatment will be discontinued early.
  For device selection, the CAP patch trauma therapy device (CAP-PTTD) will be used for lesions located on relatively flat areas of the face. In cases of lesions on areas with greater anatomical curvature (eg, the mandibular angle or near the tragus), the CAP jet trauma therapy device (CAP-JTTD) will be used in combination.
  Arms: the CAP treatment group
Device: sham CAP therapy — the device will be operated with the plasma-generating field disabled, so that no plasma will be produced. Only environmental cues such as sound will be simulated to ensure blinding.
  Arms: the placebo group
Other: standard care based on the JAAD acne guidelines — the group will receive standard care based on the JAAD acne guidelines

SUMMARY:
Acne vulgaris is a common, chronic inflammatory skin disease with complex pathogenesis and limited therapeutic options, especially for moderate-to-severe cases. Standard treatments-including topical and oral agents-are often constrained by side effects, antimicrobial resistance, and treatment resistance. Cold atmospheric plasma (CAP), a novel technology that generates reactive oxygen and nitrogen species, has demonstrated antimicrobial and tissue-regenerative properties in dermatology, but robust clinical evidence in acne management remains scarce. Existing data suggest promising efficacy and safety, yet its use in moderate-to-severe acne vulgaris has not been adequately investigated. This study aims to evaluate the efficacy and safety of two self-developed CAP devices as a potential innovative therapy for moderate-to-severe acne vulgaris.

DETAILED DESCRIPTION:
Acne vulgaris is one of the most prevalent chronic inflammatory skin diseases worldwide, with a complex and multifactorial pathogenesis. The main contributing factors include excessive proliferation of follicular keratinocytes leading to follicular plugging, dysregulated sebum production, and the overgrowth and hyperactivity of Cutibacterium acnes (formerly Propionibacterium acnes). Clinically, acne vulgaris is characterised by both non-inflammatory lesions (open and closed comedones) and inflammatory lesions (papules, pustules, and nodules), with severity ranging from mild to severe.

Current therapeutic strategies primarily target reduction of inflammation, sebum production, and microbial load. The mainstays of topical therapy are antibiotics, benzoyl peroxide, and retinoids. For moderate-to-severe cases, oral antibiotics such as minocycline and doxycycline are widely used, and oral isotretinoin remains the cornerstone for severe and refractory disease. In patients with underlying hormonal disturbances, combined oestrogen/progestin therapy may be beneficial. Nevertheless, the long-term use of systemic antibiotics is associated with potential side effects, increasing antimicrobial resistance, and limited efficacy in some patients. Isotretinoin, while highly effective, can be contraindicated or poorly tolerated due to its teratogenicity and adverse effect profile. These challenges underscore the need for innovative and alternative therapeutic approaches, particularly for patients with moderate-to-severe disease, contraindications, or treatment resistance.

Cold atmospheric plasma (CAP) has recently emerged as a novel technology in wound healing and aesthetic dermatology. CAP generates a range of reactive oxygen and nitrogen species (RONS) via glow discharge at atmospheric pressure, producing strong oxidative effects that can denature and coagulate bacterial proteins, disrupt cell membranes, and induce apoptosis of pathogenic microorganisms. In addition to its antimicrobial properties, CAP stimulates local microcirculation, enhances nutrient absorption, accelerates collagen synthesis, and promotes tissue regeneration and wound healing. CAP has been approved by the US FDA since 2008 for use in a variety of dermatological indications, including acne scars, wrinkles, superficial skin lesions, actinic keratosis, viral warts, and seborrheic keratosis. Its broad-spectrum effects offer both anti-inflammatory and skin-rejuvenating benefits, with a favourable safety profile and good patient tolerability.

Although CAP holds promise as a therapeutic modality, its application in the management of acne vulgaris, particularly moderate-to-severe cases, remains underexplored. The high cost of CAP devices and limited availability in specialised dermatology centres have restricted its widespread adoption, and robust clinical data are still lacking. In a prospective study by Wasinee et al. (Mae Fah Luang University, Thailand), weekly CAP-assisted treatment over six weeks in 31 volunteers with mild-to-moderate acne led to approximately 75% reduction in lesion count, with the greatest improvement observed in inflammatory lesions. Most adverse events were mild, including transient dryness and superficial exfoliation. Arisi et al. also reported improvements in two young patients with mild-to-moderate facial acne following CAP treatment, as assessed by lesion count, sebum output, and transepidermal water loss, with no reported adverse effects. However, data on the use of CAP for moderate-to-severe acne vulgaris-where clinical management is most challenging-are particularly scarce. To date, there have been no large, randomised controlled trials specifically evaluating CAP in this population.

Given these gaps, CAP represents a potentially innovative and adjunctive therapeutic approach for moderate-to-severe acne vulgaris, particularly in cases refractory to or unsuitable for standard treatments. In this study, we combine two self-developed CAP devices to capitalise on their respective advantages, enabling personalised and precise coverage of diverse lesion sites. This strategy aims to maximise CAP's antimicrobial and wound-healing mechanisms, and to provide robust evidence regarding its safety and efficacy in the management of moderate-to-severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years;
* Clinically diagnosed with acne vulgaris, with moderate to severe disease (Pillsbury grade III or IV, lesion count ≥50);
* Will agree to use effective contraception during the treatment period;
* Will sign a written informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Known allergy to any active component of CAP;
* Use of systemic antibiotics within 4 weeks prior to enrollment;
* Presence of dyslipidemia or other severe systemic diseases;
* Participation in other clinical trials within the past 3 months or currently enrolled in another clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
The difference in lesion clearance rate change between the CAP treatment group and the placebo group. | Baseline and up to 6 weeks after randomisation

SECONDARY OUTCOMES:
The difference between the two groups in time from randomisation to achieving 75% and 50% lesion clearance rates. | Baseline and up to 6 weeks after randomisation
The difference in change in quality of life (QoL) as measured by the QoL-acne questionnaire before and after treatment between the two groups. | Baseline and 6 weeks after randomisation

OTHER OUTCOMES:
The difference between the two groups in the incidence of the composite endpoint of erythema, edema, burning sensation, pruritus, exudation, desquamation, and scabbing. | 1 week, weeks 2-6 after randomisation, and 1, 2, and 3 months after the end of treatment
The difference between the two groups in the incidence of lesion exacerbation. | 1, 2, and 3 months after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lin Tao, MM, Principal Investigator — Shenyang Medical College; Yun-En Liu, MD, Study Chair — Shenyang Medical College
Locations (1):
- the 989th Hospital of Chinese People's Liberation Army Joint Logistic Support Force, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol